CLINICAL TRIAL: NCT00000698
Title: A Treatment Protocol for the Use of Intravenous Ganciclovir in AIDS Patients With Immediately Sight-Threatening CMV Retinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: TX 303
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 1992-04

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Retinitis; AIDS-Related Opportunistic Infections; Ganciclovir; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Retinitis; AIDS-Related Opportunistic Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency; Cytomegalovirus Infections; Acquired Immunodeficiency Syndrome | interventions — Ganciclovir

INTERVENTIONS:
Drug: Ganciclovir

SUMMARY:
To determine the safety and effectiveness of intravenous ganciclovir (also known as DHPG) in the treatment of sight-threatening cytomegalovirus (CMV) retinitis in patients with AIDS. CMV retinitis is a severe vision-threatening viral infection of the retina of the eye. It occurs in patients whose immune function has been impaired and is the most common cause of blindness in patients with AIDS. Ganciclovir (GCV) improved the signs and symptoms of CMV retinitis in approximately 80 percent of the patients treated for 2 weeks, but almost all of the patients treated with GCV had a relapse after treatment was stopped. Thus, it is important to determine if GCV can be safely given over a long period of time (maintenance therapy) and if it is effective in preventing a relapse of CMV retinitis.

DETAILED DESCRIPTION:
CMV retinitis is a severe vision-threatening viral infection of the retina of the eye. It occurs in patients whose immune function has been impaired and is the most common cause of blindness in patients with AIDS. Ganciclovir (GCV) improved the signs and symptoms of CMV retinitis in approximately 80 percent of the patients treated for 2 weeks, but almost all of the patients treated with GCV had a relapse after treatment was stopped. Thus, it is important to determine if GCV can be safely given over a long period of time (maintenance therapy) and if it is effective in preventing a relapse of CMV retinitis.

Patients are given GCV intravenously for 14 days. Then the patient receives the same dose, but only once a day, for as long as therapy is tolerated. If the retinitis worsens during the maintenance phase, the patient may again be given GCV for 14 days. Long-term treatment with GCV usually requires the surgical placement of a catheter in a large central vein in the chest or groin that is left in place indefinitely. If this is required, the procedure will be explained to the patient.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine prophylaxis for Pneumocystis carinii pneumonia.
* Topical ophthalmics.
* Topical acyclovir.

Concurrent Treatment:

Allowed:

* Hemodialysis for patients with renal impairment.

Patients must have:

* Diagnosis of AIDS and immediately sight-threatening cytomegalovirus retinitis.

Prior Medication:

Allowed:

* Zidovudine.
* Prior therapy for retinitis.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Non-immediately sight-threatening cytomegalovirus retinitis.

Concurrent Medication:

Excluded:

* Systemic investigational agents such as antimetabolites, alkylating agents, nucleoside analogs, acyclovir sodium (Zovirax).
* Interferon.
* Cytokines.
* Foscarnet (non-nucleoside pyrophosphate analog).
* Ganciclovir may be withheld for up to 21 days for an acute course with an investigational or toxic therapy or oral / IV acyclovir.

Patients with the following are excluded:

* Non-immediately sight-threatening cytomegalovirus retinitis.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Feinberg J, Study Chair
Locations (1):
- Natl Inst of Allergy & Infect Dis / Cln Ctr, Bethesda, Maryland, United States

REFERENCES:
- [Background] Feinberg J, Katz D, Mastre B, DeArmond B. Ganciclovir (GCV) in AIDS patients with immediately sight-threatening CMV retinitis (ISTCR): initial summary of "treatment IND" data. Int Conf AIDS. 1990 Jun 20-23;6(1):230 (abstract no ThB432)